CLINICAL TRIAL: NCT06838910
Title: Tislelizumab Combined With Anlotinib as Second-line Therapy in Thymoma and Thymic Carcinoma: An Open-label, Single-centre, Phase 2 Study
Brief Title: Tislelizumab Combined With Anlotinib as Second-line Therapy in Thymoma and Thymic Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-694
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-02

CONDITIONS: Thymic Carcinoma; Thymoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab + Anlotinib (Experimental)
  Interventions: Drug: Experimental: tislelizumab+anlotinib

INTERVENTIONS:
Drug: Experimental: tislelizumab+anlotinib — All patients will receive tislelizumab 200mg on Day1 every 3-week plus anlotinib 12mg or 10mg or 8mg on Day 1-14 every 3-week (Q3W) until disease progression.

SUMMARY:
It is an open-lable, single-arm, single-center, phase II clinical trial conducted in China, and plan to recruiting 20 patients who were progressed after first line chemotherapy or chemotherapy combined with immunotherapy. The purpose of this study is to evaluate the safety and efficacy of tislelizumab combined with anlotinib as second-line in thymoma and thymic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited.
2. Histologically or cytologically confirmed thymoma or thymic carcinoma.
3. Disease progression during or after first-line chemotherapy (with or without immunotherapy).
4. At least one measurable solid tumor lesion according to RECIST 1.1 criteria.
5. Estimated survival ≥ 3 months; United States Eastern Cooperative Oncology Group (ECOG) score: 0 or 1 point.
6. Vital organ function meets the following criteria:

   1. Hematological examination (no use of any blood components and cell growth factors within 14 days prior to initiation of study treatment): i. neutrophil count (ANC) ≥ 1.5×109/L; ii. platelet count (PLT) ≥100 × 109/L; iii. hemoglobin (Hb) ≥80g/L;
   2. total bilirubin (TBIL) ≤ 1.5× upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN, serum albumin (ALB) ≥28g/L;
   3. left ventricular ejection fraction (LVEF) ≥50%;
7. Female subjects of childbearing potential must have a serum pregnancy test within 7 days prior to the first dose with a negative result; and must be non-lactating; Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to comply with contraceptive requirements from the time of signing the informed consent form until 8 weeks after the end of the last treatment session.
8. Informed consent was signed.

Exclusion Criteria:

1. Prior treatment with anlotinib or any other anti-angiogenesis drugs.
2. Patients with symptomatic brain metastasis.
3. Other primary malignancy in the past 5 years, with the exception of: (radical Non-melanoma skin cancer or cured cervical in-situ carcinoma).
4. Subjects with active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis.
5. Severe infections within 4 weeks prior to inclusion.
6. Any of the following severe acute comorbidities prior to inclusion:

   1. Does not have uncontrolled pleural effusion/pericardial effusion/or ascites as determined by the investigator;
   2. Unstable angina myocardial infarction or uncontrolled congestive heart failure within 12 months;
   3. Uncontrollable hypertension;
   4. Urine routine test protein ≥++, and confirmed 24 hours urine protein> 1.0 g;
7. Imaging shows that the tumor has invaded a vital vessel perimeter or who, in the opinion of the investigator, have a high likelihood of fatal hemorrhage due to tumor invasion of a vital vessel during the follow-up study;
8. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
9. Major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to inclusion.
10. Presence of any mental disease or drug abuse disorder that may interfere with subject's ability for being compliant with study requirements.
11. Known hypersensitivity or allergy to monoclonal antibody.
12. Is receiving systemic steroid therapy < 2 weeks prior to the first dose of trial treatment or receiving any other form of immunosuppressive medication.
13. Diagnosis of immunodeficiency or undergoing systemic glucocorticoid therapy or any other immunosuppressive therapy that was continued within 2 weeks prior to the first dose.
14. Participation in another clinical trial within 28 days.
15. Any condition that, in the opinion of the investigator, would interfere with evaluation or interpretation of patient safety or study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Two years of observation after enrollment
  Objective Response Rate (ORR) refers to the proportion of patients whose cancer shrinks (partial response) or disappears (complete response) after treatment.

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years of observation after enrollment
  The time from enrollment to death due to any reason.
Progression free survival (PFS) | Two year of observation after enrollment
  The time from the beginning of randomization to the progression of tumor development or death for any reason.
Duration of response (DOR) | 24 months
  DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No